CLINICAL TRIAL: NCT05164172
Title: Long-term, Open-label (Dose-blinded), Extension Study of Eptinezumab in Children and Adolescents With Chronic or Episodic Migraine
Brief Title: A Study With Eptinezumab in Children and Adolescents (6 to 17 Years) With Chronic or Episodic Migraine
Acronym: REJOIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19379A; 2022-502917-27-00 (Other: EU CTR No.)
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eptinezumab 300 mg (Experimental): Participants will receive 3 intravenous (IV) infusions of eptinezumab 300 mg (weight adjusted) at Weeks 0, 12, and 24.
  Interventions: Drug: Eptinezumab
- Eptinezumab 100 mg (Experimental): Participants will receive 3 IV infusions of eptinezumab 100 mg (weight adjusted) at Weeks 0, 12, and 24.
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Concentrate for solution for infusion
  Other Names: Vyepti

SUMMARY:
The main goal of the study is to assess the long-term safety of eptinezumab on children and adolescents ages 6 to 17 with chronic or episodic migraine.

DETAILED DESCRIPTION:
This is an extension study for participants aged 6 to 17 with migraine who completed either studies 19356A (NCT04965675) (chronic migraine [CM] study in adolescents) or 19357A (episodic migraine [EM] study in children and adolescents). All participants who complete the Week 12 visit of the respective lead-in study will be offered participation in this open-label extension (OLE) study, unless there is a safety concern precluding a participant's participation in the study. Participants originally randomized to 100 milligrams (mg) (weight adjusted) in the double-blind lead-in study (Study 19356A or Study 19357A) will continue on the same dose (100 mg, weight adjusted) in the OLE study. Participants randomized to the 300 mg dose (weight adjusted) in the double-blind lead-in study will continue on 300 mg (weight adjusted) in the OLE study. Participants who were assigned to placebo in the double-blind lead-in study will be randomly allocated to one of the two treatment groups: eptinezumab 100 mg (weight adjusted) or eptinezumab 300 mg (weight adjusted) with a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

- The participant must have completed Week12 (completion) visit of either Study19356A (CM) or Study19357A (EM) immediately prior to enrolment into this OLE study.

Exclusion Criteria:

* The participant has an adverse event or other safety concerns that are deemed related to double-blind treatment received in the lead-in study and is considered a potential safety risk by the investigator.
* During lead-in Study19356A or Study19357A:
* participant experienced ananaphylactic reaction or another severe and/or serious hypersensitivity reaction to the investigational medicinal product (IMP) infusion, as assessed by the investigator
* the participant had a serum alanine aminotransferase (ALT) or aspartate aminotransferase(AST) value >5 times the upper limit of the reference range that was confirmed by testing <2 weeks later.
* the participant had a serum ALT or AST value >3times the upper limit of the reference range and a serum total bilirubin value >2times the upper limit of the reference range.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events | Baseline up to Week 44

SECONDARY OUTCOMES:
Free Eptinezumab Plasma Concentration | Baseline, Weeks 8, 12, 24, 36, and 44
Number of Participants With Specific Anti-Eptinezumab Antibodies (Anti-Drug Antibodies [ADA]) | Baseline (Week 0), Weeks 8, 12, 24, 36, and 44
Number of Participants With Specific Anti-Eptinezumab Antibodies for Neutralizing Activity (NAb) | Baseline (Week 0), Weeks 8, 12, 24, 36, and 44
Change From Baseline in Pediatric Migraine Disability Assessment Questionnaire (PedMIDAS) Score at Weeks 12, 24, and 36 | Baseline, Weeks 12, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (67):
- United States (19):
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - A G A Clinical Trials, Hialeah, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - University of South Florida, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Michigan State University - Department of Neurology, East Lansing, Michigan
  - Helen Devos Childrens' Hospital - PIN, Grand Rapids, Michigan
  - Dent Neurosciences Research Center Incorporated, Amherst, New York
  - True North Neurology, Commack, New York
  - OnSite Clinical Solutions, LLC - Randolph Rd - Charlotte, Charlotte, North Carolina
  - Childrens Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - Road Runner Research Ltd, San Antonio, Texas
  - Children's Specialty Group - 3 Commercial Place, Norfolk, Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - Children's Wisconsin - Milwaukee Campus - PIN, Milwaukee, Wisconsin
- Argentina (6):
  - Hospital Privado de La Comunidad, Mar del Plata, Buenos Aires
  - Expertia S.A- Mautalén Salud e Investigación, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital de Niños de La Santisima Trinidad, Córdoba-Barrio Crisol, Córdoba Province
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
- Canada (3):
  - Vancouver Island Health Authority, Victoria, British Columbia
  - The Kids Clinic, Ajax, Ontario
  - London Health Sciences Centre -800 Commissioners Rd E, London, Ontario
- Italy (8):
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - INCIPIT - PIN, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - AO Brotzu - Clinica di Neuropsichiatria dell'Infanzia e dell'Adolescenza - INCIPIT - PIN, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa, Tuscany
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia
- Mexico (4):
  - Centro de Investigacion Medico Biologica y de Terapia Avanzada S.C., Guadalajara, Jalisco
  - Clinical Research Institute SC-Mexico, Ampl San Lucas Tepetlacalco, México
  - ICARO Investigaciones en Medicina, S.A de C.V, Chihuahua City
  - Instituto de Investigationes Clinicas para la Salud A.C., Durango
- Poland (6):
  - Centrum Medyczne Plejady Magdalena Celinska - Lowenhoff, Michal Zolnowski Spolka komandytowa, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim, Lesser Poland Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw, Lower Silesian Voivodeship
  - ETG Lublin - PPDS, Lublin, Lublin Voivodeship
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - ETG Neuroscience - PPDS, Warsaw, Masovian Voivodeship
- Portugal (5):
  - ULS de Almada-Seixal, EPE - Hospital Garcia de Orta, Almada, Setúbal District
  - ULS de Santo António, EPE - Centro Materno Infantil Norte, Porto Covo, Setúbal District
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospital Pediátrico de Coimbra, Coimbra
  - ULS de São João, EPE - Hospital de São João, Porto
- Serbia (5):
  - Childrens University Hospital, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Children and Youth Health Care Institute of Vojvodina, Novi Sad
  - Clinical Centre of Vojvodina, Novi Sad
- Spain (5):
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Turkey (Türkiye) (2):
  - Eskisehir Osmangazi Universitesi Tip Fakultesi Hastanesi, Eskişehir
  - Mersin University Medical Faculty, Mersin
- United Kingdom (4):
  - Great Ormond Street Hospital - PPDS, London, London, City of
  - Royal Hospital for Children and Young People - PIN, Edinburgh, Midlothian
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - Queen Elizabeth University Hospital - PPDS, Glasgow